CLINICAL TRIAL: NCT05259111
Title: Acute Care at Home for Adults Undergoing Bariatric Sleeve Gastrectomy: A Randomized Controlled Trial
Brief Title: Home Hospital for Bariatric Sleeve Gastrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, David Levine, Associate Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017P002583e
Record Dates: First submitted 2022-02-10; First posted 2022-02-28 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Bariatric Surgery Candidate; Bariatric Sleeve Gastrectomy; Home Hospital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control, Care in the Hospital (No Intervention): After bariatric sleeve gastrectomy, patients receive their care in the hospital, as usual.
- Intervention, Care in the Home (Experimental): After bariatric sleeve gastrectomy, patients receive their care in the home.
  Interventions: Other: Home hospital

INTERVENTIONS:
Other: Home hospital — Acute care provided at home, including nurse/paramedic visits, physician visits, laboratory testing, imaging, continuous monitoring, 24/7 urgent visits, and specialty consultation.
  Arms: Intervention, Care in the Home

SUMMARY:
Providing acute care at home for medicine patients is a well-studied care model. Providing acute care at home immediately following major surgery is less well understood. The investigators seek to demonstrate the noninferiority of care at home versus the hospital for patients undergoing bariatric sleeve gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* All existing home hospital criteria apply, with the following taking precedent for this specific condition
* 21-55 years old
* Indication for bariatric laparoscopic sleeve gastrectomy per surgeon
* Caregiver capable of communicating with the home hospital team and able to stay in the same home as the patient the first night the patient is home

Exclusion Criteria:

* All existing home hospital criteria apply, with the following taking precedent for this specific condition
* Comorbidities

  * Body mass index>55
  * Chronic kidney disease
  * Heart failure
* History of

  * Chronic pain (with or without opioid use)
  * Substance use disorder
  * Venous thromboembolism
  * Stroke
  * Chronic headache
* Medications

  * Anticoagulants and anti-platelets: aspirin, clopidogrel, warfarin, and direct oral anticoagulants
  * Beta blockade
  * Immunosuppressive
  * Supplemental oxygen
* Allergy to ketorolac
* Prolonged QTc

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-02-23 (Actual); Primary Completion 2023-02-23 (Estimated); Study Completion 2023-03-23 (Estimated)

PRIMARY OUTCOMES:
Length of Stay | From day of admission to day of discharge, assessed up to 10 months
  Days spent hospitalized

SECONDARY OUTCOMES:
Motion | From day of admission to day of discharge, assessed up to 10 months
  Percent of the day lying down
Cost, direct | From day of admission to day of discharge, assessed up to 10 months
  Presented as a percentage
Opioid use | From day of admission to day of discharge, assessed up to 10 months
  Morphine milligram equivalents used

OTHER OUTCOMES:
Rate of emergency department presentation | From day of discharge to 30 days later, assessed up to 10 months
  Emergency department presentation without admission
Rate of readmission | From day of discharge to 30 days later, assessed up to 10 months
  Readmission to the hospital
BodyQ Score | From day of admission to day of discharge, assessed up to 10 months
  Sum of the following three transformed scales (total of 300 points): Satisfaction with information (100 points) + Satisfaction with doctor/surgeon (100 points) + Satisfaction with medical team (100 points)
Picker experience questionnaire - 15 | From day of admission to day of discharge, assessed up to 10 months
  0-15 points, more points better
Global experience score | From day of admission to day of discharge, assessed up to 10 months
  0-10 points, more points better
Pain score | From day of admission to day of discharge, assessed up to 10 months
  Pain score on scale of 0-10, fewer points better
Number of complications | From day of admission to day of discharge, assessed up to 10 months
  Sum of the complications included in the metabolic and bariatric surgery accreditation and quality improvement program
Bed-days saved | From day of admission to day of discharge, assessed up to 10 months
  Acute care bed days not required due to the intervention
Stage 2 diet | From day of admission to day of discharge, assessed up to 10 months
  Time to resumption of stage 2 diet, measured in hours
400mL intake | From day of admission to day of discharge, assessed up to 10 months
  Time to intake of 400mL, measured in hours
6 hours out of bed on post operative day 1 | From day of admission to day of discharge, assessed up to 10 months
  Time to 6 hours out of bed on post operative day 1, measured in hours

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Brigham and Women's Faulkner Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leff B, Burton L, Mader SL, Naughton B, Burl J, Inouye SK, Greenough WB 3rd, Guido S, Langston C, Frick KD, Steinwachs D, Burton JR. Hospital at home: feasibility and outcomes of a program to provide hospital-level care at home for acutely ill older patients. Ann Intern Med. 2005 Dec 6;143(11):798-808. doi: 10.7326/0003-4819-143-11-200512060-00008. PMID 16330791
- [Background] Levine DM, Pian J, Mahendrakumar K, Patel A, Saenz A, Schnipper JL. Hospital-Level Care at Home for Acutely Ill Adults: a Qualitative Evaluation of a Randomized Controlled Trial. J Gen Intern Med. 2021 Jul;36(7):1965-1973. doi: 10.1007/s11606-020-06416-7. Epub 2021 Jan 21. PMID 33479931
- [Background] Bryan AF, Levine DM, Tsai TC. Home Hospital for Surgery. JAMA Surg. 2021 Jul 1;156(7):679-680. doi: 10.1001/jamasurg.2021.0597. No abstract available. PMID 33909002